CLINICAL TRIAL: NCT06952543
Title: Ultrasound Perfusion Estimation for Assessment of PAD
Brief Title: Ultrasound Perfusion Estimation for Assessment of Peripheral Arterial Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Azra Alizad, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-002802; 1R01HL174785-01 (NIH)
Record Dates: First submitted 2025-04-15; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Symptomatic patients with claudication, at risk for peripheral arterial disease (PAD)
  Interventions: Diagnostic Test: Ultrasound Imaging
- Healthy Volunteers (Experimental): Healthy volunteers with normal ankle-brachial index (ABI)
  Interventions: Diagnostic Test: Ultrasound Imaging

INTERVENTIONS:
Diagnostic Test: Ultrasound Imaging — Non-invasive ultrasound will be performed using Angio Flow Reactivity Analysis (AFRA)
  The ultrasound probe will be attached to the subject's calf muscle and a pressure cuff will be secured around thigh. Ultrasound data will be collected for 1 minute.
  The cuff will then be induced to a tolerable pressure of no more than 160 mm Hg, and ultrasound data will be collected for 3 minutes while cuff is inflated.
  The cuff pressure will be released, and ultrasound data will be collected for 2 minutes after the release.
  Subject will be asked to perform 1 minute plantar flexion exercise, and ultrasound data will be collected for two minutes after the completion of exercise

SUMMARY:
The purpose of this study is to develop a new noninvasive tool for early diagnosis of Peripheral Arterial Disease (PAD) and use the proposed method for monitoring the disease progression and the response to interventional treatment in PAD patients.

ELIGIBILITY:
Inclusion Criteria:

Patient volunteers:

* Male and Female, ages 18 years old and up
* Symptom of claudication and suspected for PAD
* Scheduled for vascular testing.

Healthy volunteers:

* Male and female, ages 18-75 years old and up
* Normal BMI
* No history of smoking, cardiovascular disease, or diabetes.

Exclusion Criteria:

Patient volunteers:

* Patients with gangrene
* Patients having surgery or stent
* Patients with ulcer on their leg
* Any health condition that does not allow proper use of ultrasound scanning
* People considered in "vulnerable" populations.

Healthy volunteers:

* Include volunteers with BMI not more than 30
* No history of smoking
* No history of (diabetes, hypertension, cardiovascular diseases)
* People considered in "vulnerable" populations.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Detection of peripheral arterial disease using ultrasound perfusion estimation | Up to 4 years
  Evaluate the sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of ultrasound perfusion estimation compared to a reference standard (e.g., ankle-brachial index [ABI], CT angiography, or MR angiography) in diagnosing PAD.

SECONDARY OUTCOMES:
Detection of peripheral arterial disease longitudinal changes using ultrasound perfusion estimation | Up to 4 years
  To assess longitudinal changes in perfusion values measured via ultrasound following medical, endovascular, or surgical interventions for PAD.

CONTACTS AND LOCATIONS:
Overall Officials: Azra Alizad, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials